# DOCUMENT Informed Consent Form

OFFICIAL TITLE OF THE STUDY

Effect of Phosphoric Acid Etching Duration on the Performance of Direct Resin-Based Composite Restorations in Permanent Anterior Teeth: A Randomized Controlled Single-Center Trial

**NCT NUMBER** 

**NCT ID not yet assigned** 

SWISSETHICS REFERENCE NUMBERS

HumRes66788 | SNCTP000006373 | BASEC2025-00584

DATE OF THE DOCUMENT

**April 19, 2025** 



- University Center for Dental Medicine Basel UZB
- Mattenstrasse 40 2
- 3 CH-4058 Basel



#### Request to participate in dental research 4

- 5 Study title: Effect of Phosphoric Acid Etching Duration on the Performance
- 6 of Direct Resin-Based Composite Restorations in Permanent Anterior
- 7 Teeth: A Randomized Controlled Single-Center Trial

8 9 Layman's title: How does the etching time with phosphoric acid influence the

- 10 Behavior of tooth-colored resin fillings in anterior teeth? A clinical
- 11 Study

- 13 Dear Sir or Madam
- 14 We would like to inform you about a study on tooth-colored resin fillings for
- 15 front teeth and ask you whether you would like to take part in the examination.
- 16 tions. It is important for dentists to be aware of the effects of new interventional techniques.
- 17 methods order to further improve dental care.
- 18 We call such research a clinical trial<sup>1</sup>. In this study we want to
- 19 to find out whether the exposure time of a phosphoric acid gel has an influence on the quality of
- 20 plastic fillings on front teeth. Specifically, we would like to know whether longer or shorter
- 21 This gel has a longer application time and leads to less discoloration at the margins of the filling. This gel
- 22 is used as standard in the production of resin fillings. Until now, each
- 23 However, it is not clear how long the optimum exposure time should be. Therefore compare
- 24 In this study, we used two different application times for the gel. You need one of these
- 25 anterior filling. We would therefore like to ask you whether you would like to take part in this study.
- 26 Your participation is voluntary. The following patient information is intended to help you decide
- 27 help you with your planning. You can discuss any questions you may have about participating in the study with the investigator.
- 28 the test dentist. This is what we call the dentists who are responsible for a
- 29 study and who are responsible for you in the context of this study. If you participate
- 30 please sign the declaration of consent at the end. With your un
- 31 By signing below, you confirm that you have read and understood the patient information.
- 32 If you do not understand something, please ask the examining dentist. 33

<sup>&</sup>lt;sup>1</sup> The law uses the term "clinical trial" for this purpose.

- 34 The patient information and declaration of consent consist of four parts:
- 35 Part 1 The most important facts in brief
- 36 Part 2 This is what it's all about in detail: Information on

the study

- 37 Part 3 Data protection and insurance cover
- 38 Part 4 Declaration of consent

39

- 40 If you read **Part 1**, you will get an overview of the study.
- In Part 2, we explain the entire process and background of the study in detail.
- 42 **Part 3** contains information on data and insurance protection.
- With your signature at the end of the document, **part 4**, you confirm that you have understood everything.
- 44 and to participate.
- 45 This study was initiated by the University Center for Dental Medicine Basel UZB. This
- Institution is called the sponsor. The sponsor is responsible for, manages and finances a study program.
- 47 the.

- In the context of this study is responsible for you:
- 50 Name PD Dr. med. dent. Florin Eggmann
- 51 Address UZB, Mattenstr. 40, 4058 Basel
- 52 Telephone 061 267 26 80
- 53 079 374 13 81 (available 24 hours a day)
- 54 e-mail florin.eggmann@unibas.ch

#### 55 Part 1:

56

### The most important facts in brief

#### 57 1 Why are we this study?

- You have an anterior tooth that is missing due to caries, a defective filling or a damaged tooth.
- a tooth-colored plastic filling is required for the desired change in shape. That's why we ask
- Please indicate here whether you would like to participate in this study.
- When restoring a tooth with a resin filling, the tooth must be pre-treated.
- be applied. Pre-treatment ensures that the filling adheres well to the tooth. The pretreatment
- The standard is to treat the tooth by applying a special gel for a short time.
- 64 time on the tooth. This gel contains phosphoric acid. It is currently unclear how
- optimum exposure time of the phosphoric acid gel.
- In this clinical study, we are investigating how the duration of exposure to the phosphorus-
- acid gel the susceptibility of the fillings to marginal discoloration. Further investigated
- In this study, we examine the overall behavior of anterior fillings over time.
- This examination of the filling quality is based on a comprehensive assessment of the
- 70 fillings and the filled teeth. In **chapter 4** you will learn more about the scientific
- 71 Background to the study.

#### 72 2. what do you have to do when you take part?

- 73 Your participation in this study will last 5 years. We will visit you for 6 study visits
- 74 invite you. 5 of these 6 appointments are part of your general dental treatment
- 75 and also take place independently of your participation in the study. The other 1 appointment is a
- additional appointment and is only part of the study. Placement of the filling including documentation
- takes approx. 45-90 minutes. The first control appointment lasts 20-60 minutes. The four control appointments
- 78 mine take about 30 minutes. The number of appointments is shown in the illustration in
- 79 **Chapter 5**.
- 80 If you decide to take part, you will be randomly assigned to one of 2 groups.
- 81 They belong to either the test group or the control group. They are not wis-
- 82 to which group you belong. In the test group, you will be given the interventi-
- 83 The phosphoric acid gel is treated using a method that involves a very short exposure time
- 84 (10 seconds). In the control group, the phosphoric acid gel works longer on your tooth
- 85 (up to max. 30 seconds).
- 86 Chapter 5 provides more information on the study process and

procedure. 87

#### 3. what are the benefits and risks with participation?

89 **Benefit** 

88

- 90 You have no direct benefit from participating in the clinical trial. However, it is
- 91 It is possible that your participation will help future patients. The Nut-
- 92 The main advantage of the study is that the knowledge gained from the study
- 93 methods for the fabrication of tooth-colored resin fillings.
- 94 People who want to have their teeth colored in the future will benefit from improved treatment methods.
- 95 need a filling.
- 96 Risk
- 97 All materials used are approved and certified in Switzerland. The interventi-
- 98 The method of shortening the exposure time of the phosphoric acid gel has been proven in laboratory studies.
- 99 comprehensively examined.
- 100 Side effects may occur regardless of whether you use the intervention method or not.
- 101 the shortened exposure time of the phosphoric acid gel or the treatment method
- 102 of the control group, which involves a longer exposure time. We know
- 103 Perhaps not all the risks and side effects of the intervention method of shortening
- 104 the exposure time of the phosphoric acid gel. The following risks and side effects have been
- 105 are known in the treatment with tooth-colored resin fillings:
- 106 Hypersensitivity or pain after placement of the filling.
- 107 Chipping, fractures of the filling material and/or the adjacent tooth sub-108 stance.
- 109
- Partial or complete loss of the adhesive bond between the filling and the tooth, resulting in 110 partial or complete loss of the filling.
- 111 Air pockets in the filling material or underneath the filling
- 112 Minor, superficial injury to the gums.
- 113 Ingestion of material.
- Allergic reactions to components of the filling materials (e.g. methacrylate-114
- 115 plastics), the local anesthetic or the auxiliary parts used during the treatment.
- 116 be set.

117

118 Chapter 6 contains further information on risks and burdens.

## 120 Part 2:

122

151

## 121 This is what it's all about in detail: Information on the study

## 4 The scientific background of the study

| 123 | 4.1 Background: Why are we this study? |
|---|---|
| 124<br>125<br>126<br>127<br>128<br>129<br>130 | Adults often have front teeth that require a front tooth filling. Such an anterior filling may be necessary due to caries (a "hole in the tooth"). tooth", a defective filling that needs to be replaced, or because of a desired Change in shape of an anterior tooth. If you need an anterior filling, you get typically a tooth-colored resin filling. When placing such an artificial filling, the tooth is routinely prepared with a gel containing phosphoric acid. deals. |
| 131<br>132<br>133<br>134<br>135<br>136<br>137<br>138<br>139<br>140 | This procedure has been established for many years. There is already research in humans on Use of phosphoric acid gels when placing resin fillings. When using However, when using today's most common bonding agents ("dental adhesive"), it is It is unclear how long the optimal exposure time of the phosphoric acid gel is. Previous studies that in the laboratory have shown that the adhesive bond of the restorative material on the enamel (the outer layer of the tooth) with a shortened exposure time is the same. is as good as with a longer exposure time. In the so-called dentine, which is also called the dentin and is located underneath the enamel, the shortened exposure time of possible advantages for the adhesive bond. However, clinical studies are currently lacking to this. It is therefore currently unclear how a shorter exposure time of the phosphoric acid gel the susceptibility of the fillings to marginal discoloration. |
| 142<br>143 | In this study, we are therefore investigating whether the intervention method of a shortened onset The longer exposure time of the phosphoric acid gel just as effective as a longer exposure time. |
| 144<br>145<br>146 | All substances and materials in the study are registered in Switzerland. certified and approved. They are routinely used worldwide for tooth-colored fillings. used. |
| 147<br>148<br>149 | In this study, we are also investigating how anterior fillings as a whole over time. This examination of the filling quality is based on a comprehensive Send assessment of fillings and filled teeth. 150 |

Study information Version 2.0, 19.04.2025 Page /523

| 153<br>154<br>155 | In our study, participants are randomly divided into groups. This is important, to obtain reliable results from the study. This is called randomization. Each group receives a different treatment. There are 2 groups in our study: |
|---|---|
| 156<br>157<br>158<br>159 | <ul> <li>Group 1 (experimental group): In this group, the phosphoric acid gel is applied simultaneously to the enamel and dentin. The application time of the gel on both the enamel and the dentin is a total of 10 seconds.</li> </ul> |
| 160 | - Group 2 (control group): In this group, the phosphoric acid gel is first |
| 161 | to the enamel and only shortly afterwards to the dentin. The |
| 162 | The gel is applied to the enamel for 15-30 seconds and to the tooth surface for 10-15 seconds. |
| 163 | seconds on the dentin. |
| 164 | The study is a so-called blinded study. In this case, "blinded" means that |
| 165 | neither the participants nor the investigators know in which |
| 166 | group the participants were divided into. The practitioners who had the one- |
| 167 | However, they are not blinded, as they do not know which intervention is being used. |
| 168 | tion method. |
| 169 | The participants therefore do not know which group they belong to. And the sub |
| 170 | The examiners who evaluate the results have no knowledge of them. |
| 171 | This approach is intended to ensure that the results remain as objective as possible. |
| 172 | Randomization and blinding allow us to reliably assess how well |
| 173 | the intervention method is really effective. |
| 174 | 4. 3 Regulations on scientific research involving human subjects |
| 175<br>176<br>177 | We are conducting this study in accordance with the laws in Switzerland (Humanfor-Protection Act, data protection laws). In addition, we observe all internationally recognized guidelines. The responsible ethics committee has reviewed and approved the study. |
| 178<br>179 | Our study is a national study. The study is only being conducted at one location, the UZB, in Switzerland. |
| 180<br>181<br>182 | A description of this study can also be found on the website of the Federal Office for Health at www.kofam.ch under the SNCTP registration number or the BASEC-Number |
| 183 | |

152 4. 2 Structure of the study: How do we proceed?

| 185 | 5. 1 | What do v | ou have to | do if you | in the study? |
|-----|------|-----------|------------|-----------|---------------|

- Participation in the study is voluntary and lasts 5 years. You must adhere to the procedure
- 187 plan (→ Chapter 5.2) and also to all specifications that your dentist has issued.
- 188 dentist does.
- 189 You must inform your test dentist,
- 190 if your state of health changes, e.g. if you get worse, or
- if you have new complaints; this also applies if you discontinue the study prematurely.
- 192 (→ Chapters 5.3 and 5.4);
- 193 if you get toothache on the treated tooth or if this tooth
- 194 tooth becomes hypersensitive;
- 195 If a dentist performs a treatment on the treated study patient, he/she must tooth would like to perform;
- when you notice the loss of adhesion of the filling;
- if the filling is partially or completely lost (breaks off or becomes loose)
   detaches from the tooth);
  - if you become pregnant or are breastfeeding.
- 201 You must also note the following:
- You may not undergo dental whitening during your participation.
   have your teeth whitened. (Note: The desire for dental teeth whitening is generally not a criterion for exclusion. However, the tooth whitening at least two weeks before the resin filling is placed.
- 206 be).

#### 207 5. 2 What happens during the appointments?

- In the course of your participation, you will come to us 6 times for a study visit. 5 of these
- 209 appointments are part of your general treatment and are also paid independently of your
- 210 Study participation. The other 1 appointment is an additional appointment and includes
- 211 for the research study only. An appointment lasts about 30-45 minutes on average. The
- The sequence of dates is shown in the illustration below.
- 213 We do the following for all appointments:
- We will answer your questions.
- We will ask you guestions about your state of health.
- We examine your teeth and gums.
- We use dry ice to check whether the tooth is sensitive to cold.
- We take photos of the front teeth.

- 220 At the first appointment, we will check whether you meet the requirements for participation in the study.
- 221 fulfill. In addition, we will explain the exact process of the
- study. If you wish, you can take a few days after this appointment,
- 223 to in peace about your participation.
- 224 If you decide to take part voluntarily, you will be given the following information at the second appointment
- 225 fillings are used. We examine these fillings at the following appointments
- very precisely. In doing so, we evaluate them according to defined criteria in order to find out whether ver-
- 227 colorations occur at the edges of the fillings and how well the materials used
- 228 function.
- No data from your medical records will be used or analyzed for this study.
- 230 The following schedule shows all the necessary dates:

#### 231 Schedule: general and additional examinations

| Study<br>visit/Ter-<br>min | The current term | 1 | 2 | 3 | 4 | 5 | 6 |
|---|---|---|---|---|---|---|---|
| Approxima te duration (hours) | 0.5 | 0.75-1.5 | 0.3-1 | 0.5 | 0.5 | 0.5 | 0.5 |
| Query on<br>health<br>stood | 1 | 1 | + | 1 | 1 | ✓ | <b>√</b> |
| Assessmen<br>t of tooth<br>sensitivity | 1 | 1 | + | 1 | 1 | <b>√</b> | <b>✓</b> |
| Cold test tooth | 1 | <b>✓</b> | + | <b>✓</b> | 1 | <b>✓</b> | <b>√</b> |
| Placing dental filling | | <b>√</b> | | | | | |
| Post-<br>polishing<br>dental filling | | | (+) | | | | |
| Evaluation dental filling | | | + | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> |
| Photos tooth | | <b>√</b> | + | ✓ | ✓ | <b>√</b> | <b>√</b> |

| 233 | | |
|---|---|---|
| 234<br>235<br>236<br>237 | The schedule on the previous page shows all dates. The <b>general examinations courses</b> are with a <b>tick</b> (✓). The <b>additional study-specific un examinations</b> are <b>with a plus sign</b> (+). Only these studies represent therefore represent an additional expense for you. | |
| 238<br>239<br>240 | about the da | the appointments together with you. You receive a precise overview ates. We kindly ask you to inform us quickly if you still need to make an appointment. ant reasons. |
| 241 | 5. 3 | When does participation in the study end? |
| 242 | For you, pa | rticipation lasts 5 years and ends after the 6th date. You can choose your part |
| 243<br>244<br>245 | you no long | o stop taking the program earlier at any time (→ Chapter 5.4). You do not have to explain why er wish to participate. If you would like to end your participation earlier yourself any questions, please speak to your investigator. |
| 246 | If you end y | our participation prematurely, this has no influence on your further dental treatment. |
| 247<br>248 | | e and treatment (→ Chapter 5.4 for alternative treatment options). case, we will carry out a final examination for your safety. |
| <ul><li>249</li><li>250</li><li>251</li><li>252</li><li>253</li><li>254</li></ul> | If you discontinue the study earlier please contact your investigator // your investigator's dentist continue to inform you if your state of health changes, e.g. if you feel unwell. you feel worse or if you have new complaints. If your participation is premature ends, we will retain the data collected up to that point (e.g. information on the status of the payer). and the filling and photographs of the tooth with the filling) are still available for the study. evaluate. Your study data and samples will remain encrypted (→ Chapter 9). | |
| 255<br>256<br>257 | for example | o have to ask you to end the study early. This is if you want to use a material that is used for the fabrication of tooth-colored in the study. |
| 258 | 5. 4 | What happens if you do not wish to participate? |
| 259<br>260<br>261<br>262 | Even if you are not part in this study, we will treat and care for you dentally. medical treatment in accordance with current standards. If you do not take part in the study If you would like to take part in a clinical trial, your dentist will advise you on alternative options. treatment options. | |
| 263 | 5. 5 | Pregnancy |
| 264<br>265 | Except in emergencies, pregnant and breastfeeding women are generally not allowed to eat. of fillings. | |
| 266<br>267 | For women who may become pregnant: At the time of the filling placement, you may not be pregnant. We will therefore provide you with a pregnancy test, | |

| 268<br>269 | to be able to rule out pregnancy. In addition, at the time of the filling placement. 270 |
|---|---|
| <ul><li>271</li><li>272</li><li>273</li></ul> | If pregnancy or breastfeeding occurs during the follow-up period participation in the study is still possible. In this case, the dates can be for the follow-up examinations, which only include a short dental check-up, after consultation with the dentist. |
| 274 | The dosage can be adjusted in consultation with you and according to your doctor's recommendation. |
| 275 | You will discuss these questions with your examining dentist. 276 |
| 277 | 6 Risks, burdens and side effects |
| 278 | 6.1 What risks and stresses can occur? |
| 279<br>280<br>281<br>282<br>283<br>284 | There are risks and burdens involved in participating in this study, as with any medical study. treatment. Some risks are already known, others are still unknown. These Uncertainty is not unusual in the context of studies. In <b>chapter 6.2</b> you will find a List of the most common and most serious risks. Many side effects are (dental) medical treatable. During the study, we will inform you about all new findings on risks and treatment options. and side effects. |
| 285<br>286 | With a new intervention method, it is possible that there are risks that we have not yet identified. know. |
| 287<br>288<br>289<br>290<br>291<br>292 | To date, there have been no studies in the dental literature on the effects of The shorter exposure time of phosphoric acid gel has a positive effect. However, the dental adhesion promoters that we use, also for application without prior use of Phosphoric acid approved. Especially for fillings in the cervical area and fillings in Many dentists use these bonding agents without phos- phosphoric acid gel. This indicates that the shortened exposure time of the phosphoric acid |

294

295

296

gel is highly unlikely to pose any serious risks.

List of these risks of the investigations. 297

In addition, there are risks associated with the medical examinations that we are investigating in this

do. You will already be familiar with some of the tests. In chapter 6.3 you will find a

Here you will find information about the most common and most serious side effects, that we already know.

#### We use the following descriptions for this:

| very often | We find the side effect in more than 10 people out of 100 (more than 10%). |
|---|---|
| frequently | We find the side effect in 1 to 10 people out of 100 (1%-10%). |
| occasionally | We find the side effect in 1 to 10 people out of 1,000 (0.1%-1%). |
| rare | We find the side effect in 1 to 10 people out of 10,000 (0.01%-0.1%). |
| very rare | We find the side effect in less than 1 person in 10,000 (less than 0.01%). |

303

304

305

306

307

308 309

310 312

313

314

315

316

317

318

319

320

321

322

323

324

325

#### Common side effects are:

- Hypersensitivity or pain after placement of the filling.
  - o Consequences: Depending on the degree of severity, the course of the disease will be described in additional

The patient is observed at regular intervals or an intervention required. If required a painkiller that you tolerate well. If strong
If pain occurs, the filling is replaced or an additional

If pain occurs, the filling is replaced or an additional

root canal treatment. 311

#### Occasional side effects are:

- Chipping, fractures of the filling material and/or the adjacent tooth substance.
  - o Consequences: The filling must repaired or replaced.
- Partial or complete loss of the adhesive bond between filling and tooth, resulting in partial or complete loss of the filling.
  - o Consequences: The filling must be repaired or replaced.
- Air pockets in the filling material or underneath the filling
  - Consequences: Depending on the location and size of the air pocket, the filling repaired or replaced.
- Minor, superficial injury to the gums
  - Consequences: Such injuries usually do not require treatment and on their own within about 1-2 weeks. If required You can use a wound ointment that you can apply to the gums and/or a Mouthwash solution that supports healing. 327

326 328 329

330

331

332

334

335

336

337

#### Rare side effects are:

- Ingestion of material.
  - Consequences: Ingestion does not usually lead to any problems, as no side effects are to be expected due to the small quantities. 333

Very rare side effects are:

- Allergic reactions to components of the filling materials (e.g. Methacrylate plastics), the local anesthetic or the auxiliary parts used in the treatment. can be used.

| 338 | <ul> <li>Consequences: Patients with known or suspected allergies to</li> </ul> |
|---|---|
| 339 | These substances are excluded from treatment with such materials. |
| 340 | closed. Nevertheless, despite these precautionary measures, in rare cases |
| 341 | severe allergic reactions, such as anaphylactic shock, can occur. |
| 342 | shock, which require immediate emergency treatment. |

| 343<br>344 | 6. 3 | Risks and burd | lens from exam | ninations in the | stu- | |
|---|---|---|---|---|---|---|
| 345<br>346<br>347<br>348 | 5.2). These 6 | ve a negative impact | d and tested proce | edures. Nevertheles | s, they can involve risks<br>y there are the following | |
| 349 | - 1 | Brief pain stimulus du | ue to the cold test | on the tooth | | |
| 350 | - 1 | Additional examinatio | n date | | | |
| 351 | 7 Financing | and compensation | | _ | _ | |
| 352<br>353<br>354<br>355 | paid by the c | ent AG will provide y | dent AG. The filling | g materials and sele | e UZB and the ected instruments for g and polishing the fillin | igs free of |
| 356<br>357 | The research conduct of the | | o direct financial be | enefit from the imple | ementation of the projec | t. |
| 358<br>359<br>360 | to cover the | Payment can be ma | ccording to the usi | ual fee model for de | yourself. Intal treatment in the Ithe insurance compan | y or |
| 361 | Depending of | n the individual circu | mstances. | | | |
| 362<br>363<br>364<br>365 | is necessary<br>You will rece | and is not of the reg | gular check-up app | pointments, the patie | s used to assess the strent receives a I be charged according | |
| 366<br>367 | | ne travel costs for the 50.00 for 2nd class | | pointment after the | placement | |
| 368<br>369<br>370 | | | | | the not for financial compe | ensation. |
| 371 | 8. results fro | om the study | | | | |
| 372<br>373<br>374<br>375 | Your test der<br>that are not i | <u>-</u> | also incidental find changes to the ora | ings. Incidental find<br>al mucosa, for exam | to you by your dentist.<br>ings are "concomitant r<br>iple. We | |
| 376<br>377 | • | t know and which we | | vill also inform you v | vhich you are aware.<br>vhen we have a<br>Page /1: | 323 |

| 378 | Find the risk of a disease that can be prevented by taking preventive measures. |
|---|---|
| 379 | can. If you do not wish to be informed, please discuss this with your dentist. |
| 380 | your examining dentist. Some incidental findings are always reported, for example, |
| 381 | if other persons are endangered or if it must be reported by law. |
| 382 | There are also the overall results of the study, which are based on the data from all participants |
| 383 | come. This includes, for example, knowing more about the behavior of the front |
| 384<br>385 | dental fillings over time (→ Chapter 4.1). These results will affect you and your health directly. At the end of the study, your investigator dentist will give you |
| 386 | but would be happy to send you a summary of the overall results of the study if you wish. |
| 387 | the results. In addition, the results are presented in layman's terms after the end of the study. |
| 388 | Language published (link or reference, expected from 2031), 389 |

## 390 Part 3:

## 391 Data protection and insurance cover

| 392 | 9. Protection of data |
|---|---|
| 002 | |
| 393<br>394<br>395 | We protect your data (e.g. information on the condition of your teeth and other dental data). information from your medical history). For the protection of data, the Switzerland has strict legal regulations. |
| 396<br>397<br>398<br>399<br>400 | The Swiss Data Protection Act gives you the right to information, rectification and Receipt of your data that is collected, processed and forwarded as part of the study. These rights may be exercised in exceptional cases due to other legal or regulatory requirements. requirements cannot always be guaranteed. If you have any questions, please contact please contact your test. |
| 401 | 9.1 Encryption of data |
| 402<br>403<br>404<br>405<br>406<br>407<br>408<br>409<br>410<br>411 | Each study generates data from the investigations (e.g. information on the condition of the teeth and the filling). This data is documented. This is usually done electronically in large tables, the so-called "data collection sheets". All data is documented in encrypted form. "Encrypted" means that personal information that you directly identifiable are stored <i>separately</i> from the test results. the. For this purpose, there is a list (key list) that each person is assigned a unique code. identified. For example, your name, date of birth or place of residence are <i>not</i> directly listed in the database. data collection form. This key list remains at the institute for a period of 20 years. UZB and is then destroyed. No one else receives this key list. Special exceptions are regulated in chapter 9.5. |
| 412<br>413<br>414<br>415 | If we pass on data for the purpose of this study - to other professionals or organizations - we will not be able to use it. organizations that carry out further investigations - then the data is always encrypted. and your personal data is protected. This also applies if the data is transferred abroad. be passed on. |
| 416 | |

| 417 | 9. 2 | Safe handling of data during the study |
|---|---|---|
| 418<br>419<br>420<br>421<br>422 | Study. He is must compli | UZB is responsible for the secure handling of your data from this responsible for ensuring that the applicable laws, e.g. data protection laws, ed with. This also applies if (encrypted) data is used for investigations in other countries. rotection laws less favorable. This is how the sponsor protects his study: |
| 423<br>424<br>425<br>426<br>427<br>428<br>429<br>430<br>431<br>432<br>433 | in an encryptifilling quality on a server gums and the folder. Only to OneDrive, a stored in a side centers arou and Australia access your Sometimes in | your data is recorded and transmitted electronically. The data is stored in ed form on an ISO-certified server in the Netherlands (data and a backup copy of this data on an ISO-certified storage medium. In Ireland. The image data (photographs that exclusively show the teeth, see oral mucosa) are located in a password-protected the study team has access to it. They are stored in Microsoft secure cloud storage service. The image data is not only stored in a ngle location, but on several servers in different Microsoft repositories. Indit the world - including in North America, South America, Europe, Asia and Nevertheless, there is always a certain residual risk that strangers may be on personal data (e.g. risk of "hacking"). |
| 435<br>436<br>437 | • | ator dentist. This also applies to other doctors who giving your consent at the end of the document, you authorize this. Secure handling of data after the end of the study |
| 438<br>439<br>440 | Your data. T | remains responsible for the safe handling of the study after the end of the study. ne law stipulates that all study documents, e.g. the data collection luding the data sheets, stored for at least 20 years. |
| 441<br>442<br>443 | | this long period, study data remains encrypted. Health-relevant data cal history, including from this study, are and remain important for your treatment. ssible. |
| 444<br>445<br>446<br>447<br>448 | The results a<br>Your encrypt<br>However, da | whas been completed, the results are usually published in scientific journals. In published. The results are also reviewed by other experts. In ed data must be forwarded to these specialists. The ta may not used for new research purposes. Therefore the your separate consent (→ Chapter 9.4). |
| 449<br>450 | 9. 4 | Further use and disclosure of your data in other, future studies |
| 451<br>452<br>453 | used for this | om this study is very important for future research. Data which experiment can possibly be used for other experiments. passed on (also abroad). |

| 454<br>455<br>456<br>457 | Please read the additional declaration of consent at the end of the document carefully by. Please sign the consent form if you wish to carry out further research with your data. in the future. Even if you do not agree, you can still in the study. | |
|---|---|---|
| 458 | 9. 5 | Inspection rights during inspections |
| 459<br>460<br>461 | The implementation of this study can be verified. The review is carried out by authorities such as the responsible ethics committee. The sponsor must also carry out such reviews. to the quality of this study and the results. | |
| 462<br>463<br>464<br>465 | For this purpose, a small number of specially trained people are given insight into your personal data and your medical history. The data is therefore <i>not</i> required for this review. encrypted. The people who see your unencrypted data are subject to confidentiality. obligation. | |
| 466 | As a study ¡ | participant, you have the right to view your data at any time. 467 |

## 468 10. insurance cover

| nt of damage attributable to an approved and medically standardized |
|---|
| product / medical device or are also attributable to the use of a standard |
| ould have occurred, the same liability rules apply as in the case of treatment |
| a study. In such a case, the liability insurance of the |
| costs / compensation. |
| f |

#### 475 Part 4:

## 476 Declarations of consent

- 477 This consent consists of two independent declarations of consent:
- Informed consent for participation in this study Effect of Phosphoric Acid Etching
   Duration on the Performance of Direct Res-in-Based Composite Restorations in Permanent Anterior Teeth: A Randomized Controlled Single-Center Trial
- Declaration of consent for the further use and disclosure of data from this
   Study in coded form for further research.
- Please read this form carefully. Please ask us if there is anything you do not or if there is anything else you would like to know. To participate, your written
- 485 Consent required.

#### 486 Declaration of consent to participate in the study

| BASEC number | |
|---|---|
| Title of the study | Effect of Phosphoric Acid Etching Duration on the Performance of Direct Res-in-Based Composite Restorations in Permanent Anterior Teeth: A Randomized Controlled Single-Center Trial |
| Layman-understandable title | How does the etching time with phosphoric acid influence the behavior of tooth-colored resin fillings in anterior teeth? A clinical study |
| Responsible institution (Sponsor with address) | University Center for Dental Medicine Basel UZB Mattenstrasse 40 CH-4058 Basel |
| Place of implementation | University Center for Dental Medicine Basel UZB Mattenstrasse 40 CH-4058 Basel |
| Examining dentist at the place of study | PD Dr. med. dent. Florin Eggmann |
| :<br>Surname and first name in block capitals: Date of<br>birth: | |

487 I have received verbal and written information about the study, namely 488 by the test dentist who signs below. 489 490 The investigator has explained to me the purpose, procedure and risks of the 491 study and the treatment method. 492 493 I am taking in the study voluntarily. 494 495 The examining dentist has explained to me which standard treatments are possible. 496 there are outside the study. 497 498 I had enough time to this decision. I keep the written in 499 formation and receive a copy of my written declaration of consent. 500 501 I can end my participation at any time. I don't have to explain why. Also 502 if I stop participating, I will continue to receive my medical treatment. 503 The data up to this point will be analyzed as part of the study. 504 valued. 505 506 If I resign, the data remains encrypted. 507 508 If it better for my health, the examining dentist can give me the following information 509 doctor the study at any time. 510 I understand that my data will only be forwarded in encrypted form for this study. 511 512 are sent abroad. The sponsor shall ensure that the data 513 protection is complied with in accordance with Swiss standards. 514 515 In case of results // In case of results and/or incidental findings that directly affect my health 516 I will be informed of any changes that affect my health. If I do not wish to be informed, I discuss this with 517 my test . 518 519 My general practitioner may use data from my medical history that is required for the study. 520 that are important the investigator. This also applies to an-521 other doctors who treat me. 522 523 The responsible experts of the sponsor, the Ethics Committee and the Drug 524 Swissmedic may view my unencrypted data for inspection. All 525 these persons are subject to a duty of confidentiality. 526 The liability insurance of the institution UZB insures possible damages. 528 527 529

| | Place, date | Surname and first name of in block capitals |
|---|---|---|
| 530<br>531<br>532<br>533<br>534<br>535<br>536 | | Signature of participant |
| | Confirmation of the examining: I hereby confirm that I have completed the- The nature, significance and scope of the study is explained to this participant have. I confirm that I have fulfilled all obligations in connection with this study. accordance with Swiss law. Should I learn of any aspects in the course of the study, which influence the participant's willingness to take part in the study. I will her/him of this immediately. | |
| | Place, date | Surname and first name of the test in block capitals |
| | | Signature of the examining dentist |

# Declaration of consent for further use and/or disclosure of data in encrypted form

This consent does not concern you in the sense of personal participation in a study. (→ Chapter 9.4 of the patient information).

"Further use" means that your data will be stored beyond the time of your participation in the study.

and can be used in encrypted form for further research. The

can mean, for example, that examination results from you that were obtained during dental check-ups

were statistically analyzed together with a large number of other values.

or new tests are carried out with it.

547 "Disclosure" means that your data is passed on to other research persons or research institutes.

institutions in encrypted form for further research projects.

fen. These other research persons or research institutions can also be included in the training program.

country. It is the sponsor's responsibility to ensure that this country has an adequate

level of data protection comparable to that in Switzerland. 552

| BASEC number: | |
|---|---|
| Title of the study | Effect of Phosphoric Acid Etching Duration on the Performance of Direct Resin-Based Composite Restorations in Permanent Anterior Teeth: A Randomized Controlled Single-Center Trial |
| Layman-understandable title | How does the etching time with phosphoric acid influence the behavior of tooth-colored resin fillings in anterior teeth? A clinical study |
| Participant: Surname and first name in block capitals: Date of birth: | |

553

554

555 556 I authorize the use of my coded data and from this study for the (dental) meand passed on (also abroad) for further use in medical research may.

557 - I understand that the data is encrypted and the key is stored securely. 558 is maintained.

559 560

If I resign, the data remains encrypted. 561

| Place, date | Surname and first name of in block capitals |
|---|---|
| | Signature of participant |
| Confirmation of the test: I confirm that I am authorized to participate in the test. the nature, significance and scope of the further use and/or further processing of the data. of samples and/or (genetic) data. | |
| Place, date | Surname and first name of the test dentist in block capitals |
| | Signature of the examining dentist |